CLINICAL TRIAL: NCT03954964
Title: Increasing Awareness of Opioid Disposal in the Orthopedic Patient Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Christine D. Aliory, Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 18-011832
Record Dates: First submitted 2019-05-16; First posted 2019-05-17 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Knee Total Joint Replacement; Hip Total Joint Replacement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Subjects participating in a total joint class for patients undergoing planned hip and knee total joint replacement.
- Intervention Group (Experimental): Subjects participating in a total joint class for patients undergoing planned hip and knee total joint replacement will receive additional education about the disposal of opioids.
  Interventions: Behavioral: Education on disposal of opioids

INTERVENTIONS:
Behavioral: Education on disposal of opioids — Current class curriculum including education about pain management with additional education about the disposal of opioids.
  Arms: Intervention Group

SUMMARY:
Researchers are trying to determine if providing education on proper disposal of unused opioid medications to the orthopedic patient undergoing a planned hip or knee total joint replacement will increase the percentage of patients who properly dispose of unused opioids.

ELIGIBILITY:
Inclusion Criteria:

* Adult 18 + years
* Planned total hip or knee replacement surgery
* English speaking

Exclusion Criteria:

* Pediatric patients 17 and younger
* Non-English speaking patients
* Total joint replacement surgery other than Hip and Knee

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-06-03 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Disposal of unused prescription pain medication | 12 weeks post operative
  Number of subjects to self-report disposal of unused prescription pain medication on the twelve week post operative visit survey
Use of medication deactivation bag | 12 weeks post operative
  Number of subjects to self-report disposal of unused prescription pain medication via the medication deactivation bag on the twelve week post operative visit survey

CONTACTS AND LOCATIONS:
Overall Officials: Christine Aliory, APRN, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials